CLINICAL TRIAL: NCT05142943
Title: Effectiveness of Virtual Bodily Illusion Intervention in Upper Limb Motor Function, Sensibility and Pain in People With Incomplete Spinal Cord Injury.
Brief Title: Effectiveness of Virtual Bodily Illusion Intervention in Upper Limb Motor Function in People With Incomplete Spinal Cord Injury.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INV_ETICA_1681060
Record Dates: First submitted 2021-11-19; First posted 2021-12-03 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Incomplete Spinal Cord Injury; Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trail
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Visual Illusion (VI and therapeutic exercise program (EP) (Experimental): the patient will be seated in a chair with a table in front of it. The front part of the trunk will be covered with a black blanket that will be attached to the table. On the table, you will see arms and hands projected performing different types of functional manual activities that will include mobility and strength tasks. The projected arms will be adapted to the dimensions of each subject so that the patient can recognize the projected arms as theirs. This program will last 10 minutes. Then a physical exercise program for the upper extremities will be carried out:
  * General mobility and warm-up: flexion-extension joint movements, rotations, deviations, abduction-adduction, etc.
  * Gross mobility and coordination: ball games.
  * Fine mobility and coordination: writing tasks, puzzles, abacus ...
  * Strength exercises: shoulder, elbow, wrist, fingers.
  * Stretching.
  Interventions: Other: Visual illusion; Other: Physical exercise
- VI sham and EP (Sham Comparator): the configuration of the work table will be the same as in real IV, although videos of landscapes will be projected on them without any type of human or animal movement appearing on them. This program will last 10 minutes. Afterwards, a physical exercise program for the upper extremities will be carried out, detailed in Arm I.
  Interventions: Other: Physical exercise; Other: Sham Visual illusion
- VI (Experimental): only the visual illusion program will be carried out, detailed in Arm I.
  Interventions: Other: Visual illusion
- VI sham (Sham Comparator)
  Interventions: Other: Sham Visual illusion

INTERVENTIONS:
Other: Visual illusion — the patient will be seated in a chair with a table in front of it. The front part of the trunk will be covered with a black blanket that will be attached to the table. On the table, you will see arms and hands projected performing different types of functional manual activities that will include mobility and strength tasks. The projected arms will be adapted to the dimensions of each subject so that the patient can recognize the projected arms as theirs. This program will last 10 minutes.
  Arms: VI; Visual Illusion (VI and therapeutic exercise program (EP)
Other: Physical exercise — * General mobility and warm-up: flexion-extension joint movements, rotations, deviations, abduction-adduction, etc.
  * Gross mobility and coordination: ball games.
  * Fine mobility and coordination: writing tasks, puzzles, abacus ...
  * Strength exercises: shoulder, elbow, wrist, fingers.
  * Stretching.
  Arms: VI sham and EP; Visual Illusion (VI and therapeutic exercise program (EP)
Other: Sham Visual illusion — only the placebo visual illusion
  Arms: VI sham; VI sham and EP

SUMMARY:
Previous studies have shown that the neuroplasticity of the residual corticospinal fibers, the motor cortex and the spinal neurons plays an important role in the spontaneous functional recovery of people with neurological or musculoskeletal pathology. However, it is also possible to stimulate the neuroplasticity mechanisms of these structures through techniques aimed at rehabilitating different deficits (for example, motor function or sensitivity). In general, intervention programs are usually carried out, in most cases, using low-cost strategies such as therapeutic physical exercise programs.

The objective of this study is to analyze the effectiveness of visual illusion therapies in combination with conventional exercises on the symptoms and signs related to incomplete spinal cord injury that affects the upper limb.

The study will include the realization of three measurements that will be carried out one day before starting the program, one day after finishing it, and one month later (follow-up).

The clinical assessment will be composed of the study of the following variables: Motor function and motor skills, Upper limb isometric force, Muscle activation, Muscle tone, Quality of life, Functionality. All interventions will last eight weeks and will be planned according to the availability of volunteers. In each session, it will be recorded if any type of adverse effect occurs. There will be four types of interventions: i. Visual Illusion (IV) and therapeutic exercise program (PE), ii.placebo and PE, iii. IV, iv. IV placebo.

DETAILED DESCRIPTION:
Approximately 60% of people with a spinal cord injury have an incomplete injury. This causes alterations in strength, sensitivity, and muscle tone, which leads to a marked loss of functionality. This supposes a profound psychological and socioeconomic impact on the life of the affected person, in addition to the implicit physical impact.

After an injury of this type, there is a spontaneous functional recovery that may have a different path depending on the characteristics of the injury and the person. Previous studies have shown that the neuroplasticity of the residual corticospinal fibers, the motor cortex, and the spinal neurons play an important role in the spontaneous functional recovery of people with neurological or musculoskeletal pathology. However, it is also possible to stimulate the neuroplasticity mechanisms of these structures through techniques aimed at rehabilitating different deficits (for example, motor function or sensitivity). In general, intervention programs are usually carried out, in most cases, using low-cost strategies such as therapeutic physical exercise programs.

This nervous reorganization and recovery can also be influenced by the activity of mirror neurons, which are found in motor and premotor areas and also in other cortical and subcortical areas; and they report activation when they observe an action with a specific purpose. The activity of these neurons has been studied in different populations with involvement of the nervous and musculoskeletal system, such as cerebrovascular accidents, head injuries, Parkinson's, Alzheimer's, or carpal tunnel syndrome. For its study, experimental investigations have been carried out applying different interventions that modify the activity of mirror neurons, such as mirror therapy, virtual reality therapies, or Action-Observation therapies. Of these, in general, promising results have been obtained in all these populations, except in the case of Alzheimer's disease in an advanced stage.

However, these treatments have not been investigated in the recovery of the upper limb in people with incomplete spinal cord injury.

For all the above, the objective of this study is to analyze the effectiveness of visual illusion therapies in combination with conventional exercises on the symptoms and signs related to different pathologies of the nervous and musculoskeletal systems that affect the upper limb. Specifically, it is intended to know the impact of visual illusion therapy on:

* The motor function of the arm and hand.
* The functionality.
* The isometric strength of the upper extremities.
* Muscle tone, rigidity, and elasticity of the muscles of the arms.
* Neuropathic pain.
* The fine motor skills of the hand.
* The upper limb functionality.

Therefore, this study aims to provide knowledge to the scientific community on how neuroplasticity mechanisms and specifically mirror neurons can influence the rehabilitation of people with incomplete spinal cord injury and, in addition, propose a specific treatment methodology for the rehabilitation of the upper extremities in this type of population.

All procedures will be carried out under the principles of the Declaration of Helsinki (World Medical Association) and will be approved by the ethics committee of the University of Valencia. In addition, all participants will be asked to sign an informed consent that will include all the sections required by this committee.

A minimum of 20 participants per group is established, establishing a power of 80%, an ability to detect a small effect size (Coehn's d = 0.3) for the main variable mobility measured with Nedcodo Agile and a probability of type I error. of 0.05, resulting in a total of 80 participants. In order to minimize possible losses, 25% more patients will be added per group, so 100 people will participate in the study.

The study will include the realization of three measurements that will be carried out one day before starting the program, one day after finishing it, and one month later (follow-up). These will be carried out by team members who are blind to the assignment of the interventions. In the first evaluation, anthropometric and demographic data (i.e. height, weight, age, educational level, possible comorbidities, etc.) will be collected in order to control, in case of heterogeneity, these confounding variables.

The data analysis will be carried out using the SPSS statistical program (version 26). The normality of the sample will be analyzed using the Shapiro Wilk test and homoscedasticity using the Levene test. For the comparison between groups, a mixed factorial ANOVA will be used, and for the comparison between pairs of groups the Bonferroni correction will be used. In the event that there may be a confounding factor that meets the requirements to be analyzed as a covariate, an ANCOVA will be used. Statistically significant differences will be assumed when the p-value is less than 0.05.

All interventions will last eight weeks and will be planned according to the availability of volunteers. In each session, it will be recorded if any type of adverse effect occurs.

There will be four types of interventions resulting of a combination of:

* Visual Illusion (IV): the patient will be seated in a chair with a table in front of it. The front part of the trunk will be covered with a black blanket that will be attached to the table. On the table, you will see arms and hands projected performing different types of functional manual activities that will include mobility and strength tasks. The projected arms will be adapted to the dimensions of each subject so that the patient can recognize the projected arms as theirs. This program will last 10 minutes.
* Therapeutic exercise program (PE): Physical exercise program for the upper extremities will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* Incomplete cervical spinal cord injury (AIS C, D or E).
* Ability to understand instructions (Mini-Mental State Examination> 23 points)

Exclusion Criteria:

* Traumatic pathology in upper limbs.
* Other alterations of the central nervous system or peripheral
* Alterations in the vestibular system.
* Concomitant diseases.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Range of motion of wrist | 7 minutes.
  Nedcodo Agile was used to assess this outcome. Nedcodo Agile is a newly developed tool by Institut de Biomecànica de València (IBV) that measures elbow and wrist range of movement in degrees of range of movement, and press force in newtons.
Range of motion of elbow | 7 minutes.
  Nedcodo Agile was used to assess this outcome. Nedcodo Agile is a newly developed tool by Institut de Biomecànica de València (IBV) that measures elbow and wrist range of movement in degrees of range of movement, and press force in newtons.
Fingers coordination. | 7 minutes.
  Hand assessment tablet app is a tool developed by Neurorehabilitation and Brain research group that assesses hand coordination and dexterity. This app counts the number of taps in a determined time and their velocity.
Rang of movement of gripper. | 7 minutes.
  Hand assessment tablet app is a tool developed by Neurorehabilitation and Brain research group that assesses hand coordination and dexterity. This app measure the range of gripper of each finger.
Graphomotricity. | 7 minutes.
  Hand assessment tablet app is a tool developed by Neurorehabilitation and Brain research group that assesses hand coordination and dexterity. This app measure the error in centimeters of graphomotricity activity.
Upper limb isometric force. | 10 minutes
  A load cell (CTCS; Mutronic) is used to assess upper limb muscles force (in Newtons).
Muscle activation. | 10 minutes.
  The BTS FreeEMG Electromyograph is used to assess upper limb muscles activation (in microV).
Severity of pain and degree of interference with feeling and function. | 5 minutes
  Brief Pain Inventory is used to assess neuropathic pain. This test measures pain severity and pain interference from 0 to 10.
Muscle tone of upper limb. Natural Oscillation Frequency. | 5 minutes
  MyotonPRO is used to assess tone or state of tension (Natural Oscillation Frequency [Hz]) of upper limb muscles.
Muscle tone of upper limb. Biomaechanical properties. | 5 minutes
  MyotonPRO is used to assess biomaechanical properties (Dynamic Stiffness [N/m], Logarithmic Decrement of natural oscillation, characterizing and Elasticity) of upper limb muscles.
Muscle tone of upper limb. Viscoelastic properties | 5 minutes
  MyotonPRO is used to assess viscoelastic properties (Mechanical Stress Relaxation Time [ms], Ratio of deformation and Relaxation time, characterising Creep (Deborah number)) of upper limb muscles.
Spasticity of upper limb | 2 minutes
  Modified Ashworth Scale (from 1 to 4):
  0: No increase in muscle tone.
  1: Slight increase in muscle tone, with a catch and release or minimal resistance at the end of the range of motion when an affected part(s) is moved in flexion or extension.
  1+: Slight increase in muscle tone, manifested as a catch, followed by minimal resistance through the remainder (less than half) of the range of motion.
  2: A marked increase in muscle tone throughout most of the range of motion, but affected part(s) are still easily moved.
  3: Considerable increase in muscle tone, passive movement difficult. 4: Affected part(s) rigid in flexion or extension..

SECONDARY OUTCOMES:
Quality of life index- Spinal cord injury | 8 minutes
  Total quality of life score, health and functioning subscale, social and economic subscale, psychological/spiritual subscale, and family subscale. The scales (satisfaction and importance) are on a 6-point Likert scale, ranging from 1, very dissatisfied (very unimportant), to 6, very satisfied (very important). Five scores are generated (i.e. total and 4 domains) on a 0 - 30 scale.
Independence | 5 minutes
  The spinal cord independence measure (SCIM) was used. Scores range from 0-100, where a score of 0 defines total dependence and a score of 100 is indicative of complete independence. Each subscale score is evaluated within the 100-point scale (self-care: 0-20; respiration and sphincter management: 0-40; mobility: 0-40).
Press force (Newtons) | 7 minutes
  Nedcodo Agile was used to assess this outcome. Nedcodo Agile is a newly developed tool by Institut de Biomecànica de València (IBV) that measures elbow and wrist range of movement in degrees of range of movement, and press force in newtons.
Propioception | 5 minutes
  Hand assessment tablet app is a tool developed by Neurorehabilitation and Brain research group that assesses hand coordination and dexterity. This app measure the error in centimeters of graphomotricity activity with close eyes, reproducing an exercise pretrained.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultat de Fisioteràpia, Universitat de València, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No